CLINICAL TRIAL: NCT03856086
Title: The Impact of Caregiver Distress Screening, Targeted Referral and Consultation on MSK Caregiver, Patient and Health System Outcomes
Brief Title: Comparing Distress Screening + Consultation With Enhanced Usual Care for Caregivers of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-539
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cancer Caregivers
Keywords: Comparing Distress Screening; Consultation With Enhanced Usual Care; Supportive care; 18-539
MeSH Terms: interventions — Surveys and Questionnaires; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized between screening with the CSS-CG + consultation (S+C, and enhanced usual care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (EUC) (Active Comparator): ICs randomized to EUC following baseline questionnaire completion will be given instructions (Appendix I) on how to access or create an account to access the myMSK online portal IC Resources page (https://my.mskcc.org/login). If the caregiver does not wish to enroll in MyMSK, the research study staff will send them an email with sample referral material ( Appendix D. The IC Resources page includes links to extant MSK educational materials for ICs (e.g., "A Guide for Caregivers" [47]), contact information for psychosocial services (e.g., Caregivers Clinic in the MSK Counseling Center), and external resources (e.g., educational materials and services through the CSC, American Cancer Society, and others) (Appendix D,).
  Interventions: Behavioral: Baseline questionnaire; Behavioral: NCCN Problem List; Behavioral: FACT-GP; Behavioral: HADS
- CancerSupportSource-CG screening plus consultation (S+C) (Experimental): ICs randomized to S+C will complete the web-based CSS-CG (Appendix C) using a tablet immediately following baseline study measures. In case of technical issues, ICs may complete Appendix C with the guidance of a member of the research study team. The CSS-CG asks ICs to rate their level of concern for 33 different possible problems: if a need is rated as low (i.e., "A little" or less concern), after each problem is rated ICs will be prompted to request pertinent educational materials if they are interested. If a need is endorsed (i.e., "Moderate" or greater concern), ICs are asked through the web-based electronic platform (https://mskcc.mycarereport.com) whether they would like educational materials and/or to speak with someone about that need (i.e., receive a referral).
  Interventions: Behavioral: Baseline questionnaire; Behavioral: NCCN Problem List; Behavioral: FACT-GP; Behavioral: HADS; Behavioral: CSS-CG

INTERVENTIONS:
Behavioral: Baseline questionnaire — Baseline questionnaire on the day of the patient's surgery.
Behavioral: NCCN Problem List — NCCN Distress Thermometer
Behavioral: FACT-GP — Greater overall quality of life
Behavioral: HADS — Lower anxiety and depression
Behavioral: CSS-CG — web-based CSS-CG
  Arms: CancerSupportSource-CG screening plus consultation (S+C)

SUMMARY:
This study will help the researchers find out whether the S+C approach is better, the same as, or worse than EUC.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified caregiver to a patient receiving surgery at JRSC OR self-identified caregiver to a patient at various inpatient surgical floors (i.e., M4, M7, M8) at the Main Hospital OR self-identified caregiver to a patient at the BMT clinic.
* English fluency: Self-report by subject identifying English as the preferred language for healthcare, and self-reported degree of fluency as speaking English "Very well."
* 18 years old or older as per self report
* Agree to fulfill responsibilities as an IC during the perioperative phases as per self report

Exclusion Criteria:

* Cognitive difficulties that preclude participation in the intervention or accurate assessment in the judgment of the PI
* Medical illness that is of sufficient severity to preclude further participation in the study.
* Presenting to JRSC as the IC for a patient undergoing a prophylactic procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Number of Informal caregivers with unmet needs | 1 year
  comparing the 3-month change scores on the NCCN problem list from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Allison Applebaum, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm